CLINICAL TRIAL: NCT00000356
Title: Pharmacokinetics of LAAM in Methadone Patients
Brief Title: Evaluation of L-alpha-acetylmethadol (LAAM) in Methadone Patients - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-5; Y01-3-0012-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1992-02

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Methadyl Acetate

INTERVENTIONS:
Drug: LAAM

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of L-alpha-acetylmethadol (LAAM) in adults transferred from methadone maintenance treatment for opiate dependence.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 1991-06; Primary Completion 1992-08 (Actual); Study Completion 1992-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States